CLINICAL TRIAL: NCT05761392
Title: Precise Management System (PreMaSy) of Chronic Intractable Pain Based on a Remote and Wireless Spinal Cord Stimulation System
Brief Title: APP-based Precise Management System of Chronic Intractable Pain
Acronym: PreMaSy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Guihuai Wang, Director of Neurocenter of Beijing Tsinghua Changgung Hospital, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220908
Record Dates: First submitted 2023-02-09; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Pain, Chronic; Pain, Intractable
Keywords: Pain management; Spinal cord stimulation; Remote programming; Mobile health
MeSH Terms: conditions — Chronic Pain; Pain, Intractable; Agnosia

STUDY DESIGN:
Intervention Model Description: After taking the stimulator implantation surgery, participants in the interventional group are asked to take conventional follow-up including 1-, 3-, 6-month post-operative. Other than that, participants will be asked to take additional self-assessments, including daily pain state and monthly health conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precise management (Experimental): Participants will be asked to take daily pain state and monthly health condition assessments.
  A warning for the physicians will be given when participants reach daily assessment threshold. Remote interventional meeting will be scheduled and stimulation parameters will be adjusted accordingly.
  Participants will also be asked to take conventional follow-up at 1-, 3-, and 6-month post-operative.
  Interventions: Other: Precise management
- Conventional management (No Intervention): Participants will be only asked to take conventional follow-ups at 1-, 3-, and 6-month post-operative. During these follow-ups, they will be asked to score VAS based on general pain state, and take questionnaires including EQ-5D-5L, PSQI, PGIC, CGI-I.

INTERVENTIONS:
Other: Precise management — The daily pain state assessments contain three components, the visual analogue scale (VAS) based on pain intensity, time-intensity curve throughout the day, and pain locations. The VAS scores from the first seven post-operative days will be collected as the baseline data. The interventional threshold will be determined by adding 30 mm (if the scale length were 100 mm) to the baseline mean. If participants score above the threshold three times in a row, a warning will be sent to their physicians. A remote meeting will be scheduled and stimulation settings will be adjusted accordingly.
  Arms: Precise management

SUMMARY:
The goal of this clinical trial is to learn about a new management system in chronic and stubborn pain patients who accept therapy of spinal cord stimulation (SCS). Usually, these patients are required to take long-term follow-ups to ensure that the stimulator works well. The main questions it aims to answer are:

* Is it better to improve the patient's quality of life than the current conventional follow-up?
* Is it better to relieve pain in the long term than the current conventional follow-up?
* Is it possible to be applied to a large population of chronic pain patients? Participants will be randomly assigned to either a control group or an interventional group.

Participants in the control group will be given the standard SCS implantation surgery and asked to complete the conventional follow-up (at least 1-, 3-, and 6-month post-operative).

Participants in the interventional group will be given the standard SCS implantation surgery and asked to do the following things:

* Take the daily pain self-assessment questions on a mobile phone APP.
* Take the monthly healthy status self-assessment questionnaires on a mobile phone APP.
* Take the conventional follow-up (at least 1-, 3-, and 6-month post-operative). Researchers will compare the two groups to see if the life quality of the interventional group is improved.

DETAILED DESCRIPTION:
Chronic intractable pain is a disorder with complicated causes. The patient's quality of life is significantly reduced as a result of the patient's ongoing discomfort and the necessity for lengthy therapies. When patients don't respond well to medicine or other non-surgical treatments, spinal cord stimulation (SCS) is one of the surgical methods employed. The safety and effectiveness of SCS have previously been confirmed in numerous trials as a well-researched and clinically used therapy. However, the adjustment of SCS is complicated and its optimal effect relies on long-term regular follow-up. With the development of the internet, the investigators put forward a new system with remote and wireless SCS devices. Together with an exclusively developed mobile phone application, patients will be able to record their daily pain state and monthly health condition and make customized stimulation settings accordingly. This study is aimed to test the feasibility of this new precise management system. All participants will be randomly assigned to either interventional or control group. Participants in control group will be asked to take the conventional follow-up. Participants in interventional group will be additionally asked to take self-assessment on daily pain state and monthly health condition. The investigators hypothesized that this self-involved, closely monitored, and precisely adjusted system can significantly improve patients' quality of life in the long term and cut down both the financial expenses and time cost.

ELIGIBILITY:
Inclusion Criteria:

* Have been clinically diagnosed with chronic, intractable pain for more than three months.
* At enrollment, the average pain intensity is no least than 5 out of 10 cm on visual analogue scale.
* At enrollment, the age is no younger than 18-year-old.
* Ineffective or unsatisfactory conservative treatments, including but limited to: oral medication, nerve block, epidural corticosteroids, physical and psychological rehabilitation therapy, and chiropractic care.
* Voluntary to take the trial and sign the informed consent.
* Good compliance and ability to complete post-operative follow-ups.
* Basic ability to read and use a mobile phone or having a caregiver who can.

Exclusion Criteria:

* Bleeding complications or coagulation disorders.
* Mental or cognitive disorders leading to inability to complete implantation surgery or post-operative follow-up.
* Issues with spinal cord or vertebrates that are not suitable for implantation surgery.
* Systemic active infections or local infections around the surgery area.
* Pregnancy, breast-feeding, plan to be pregnant or unwilling to use contraceptive methods.
* Metastatic malignant tumors or untreated malignant tumors.
* Life expectancy of less than one year.
* Already provided with a medication pump and/or other implanted devices.
* Need for therapy or examination that must not have an implanted pulse generator (IPG), such as magnetic resonance imaging (MRI) and thermo-therapy.
* Heavily addicted to alcohol or drugs.
* VAS improvement less than 50% or stimulation intolerance during the test period.
* Unable to complete long-term online follow-ups because of hardware issues such as internet, mobile phones, and so on.
* Unwilling to participate.
* Other inappropriate situations determined by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Health Condition and Life Quality: Change From Baseline in five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) utility values at Month 1 | Baseline and Month 1
  Participants' health condition and life quality are measured by EQ-5D-5L utility values. EQ-5D-5L utility value has a minimum of 0 and a maximum of 1. Higher values mean a better health condition.
Health Condition and Life Quality: Change From Baseline in five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) utility values at Month 3 | Baseline and Month 3
  Participants' health condition and life quality are measured by EQ-5D-5L utility values. EQ-5D-5L utility value has a minimum of 0 and a maximum of 1. Higher values mean a better health condition.
Health Condition and Life Quality: Change From Baseline in five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) utility values at Month 6 | Baseline and Month 6
  Participants' health condition and life quality are measured by EQ-5D-5L utility values. EQ-5D-5L utility value has a minimum of 0 and a maximum of 1. Higher values mean a better health condition.

SECONDARY OUTCOMES:
Pain Intensity: Change From Baseline in Visual Analogue Scale (VAS) at Month 1 | Baseline and Month 1
  Pain intensity is assessed by VAS and compared with baseline VAS score. VAS has a minimum of 0 and a maximum of 10. Higher values mean a stronger pain.
Pain Intensity: Change From Baseline in Visual Analogue Scale (VAS) at Month 3 | Baseline and Month 3
  Pain intensity is assessed by VAS and compared with baseline VAS score. VAS has a minimum of 0 and a maximum of 10. Higher values mean a stronger pain.
Pain Intensity: Change From Baseline in Visual Analogue Scale (VAS) at Month 6 | Baseline and Month 6
  Pain intensity is assessed by VAS and compared with baseline VAS score. VAS has a minimum of 0 and a maximum of 10. Higher values mean a stronger pain.
Pain Time: Change From Baseline in Time-Intensity Curve at Month 1 | Baseline and Month 1
  Temporal characteristics of pain is assessed by a time-intensity curve and compared with baseline curve.
Pain Time: Change From Baseline in Time-Intensity Curve at Month 3 | Baseline and Month 3
  Temporal characteristics of pain is assessed by a time-intensity curve and compared with baseline curve.
Pain Time: Change From Baseline in Time-Intensity Curve at Month 6 | Baseline and Month 6
  Temporal characteristics of pain is assessed by a time-intensity curve and compared with baseline curve.
Pain Location: Change From Baseline in Pain Map at Month 1 | Baseline and Month 1
  Spatial characteristics of pain is assessed by a pain map and compared with baseline pain map.
Pain Location: Change From Baseline in Pain Map at Month 3 | Baseline and Month 3
  Spatial characteristics of pain is assessed by a pain map and compared with baseline pain map.
Pain Location: Change From Baseline in Pain Map at Month 6 | Baseline and Month 6
  Spatial characteristics of pain is assessed by a pain map and compared with baseline pain map.
Health condition: Change From Baseline in EuroQol Visual Analogue Scale (EQ VAS) at Month 1 | Baseline and Month 1
  Overall health condition is assessed by EQ VAS and compared with baseline EQ VAS. EQ VAS has a minimum of 0 and a maximum of 100. Higher scores mean a better health condition.
Health condition: Change From Baseline in EuroQol Visual Analogue Scale (EQ VAS) at Month 3 | Baseline and Month 3
  Overall health condition is assessed by EQ VAS and compared with baseline EQ VAS. EQ VAS has a minimum of 0 and a maximum of 100. Higher scores mean a better health condition.
Health condition: Change From Baseline in EuroQol Visual Analogue Scale (EQ VAS) at Month 6 | Baseline and Month 6
  Overall health condition is assessed by EQ VAS and compared with baseline EQ VAS. EQ VAS has a minimum of 0 and a maximum of 100. Higher scores mean a better health condition.
Sleep Quality: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) at Month 1 | Baseline and Month 1
  Sleep quality is assessed by PSQI and compared with baseline PSQI score. PSQI score has a minimum of 0 and maximum of 21. Higher scores mean a worse sleep quality.
Sleep Quality: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) at Month 3 | Baseline and Month 3
  Sleep quality is assessed by PSQI and compared with baseline PSQI score. PSQI score has a minimum of 0 and maximum of 21. Higher scores mean a worse sleep quality.
Sleep Quality: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) at Month 6 | Baseline and Month 6
  Sleep quality is assessed by PSQI and compared with baseline PSQI score. PSQI score has a minimum of 0 and maximum of 21. Higher scores mean a worse sleep quality.
Global impression: Change From Baseline in Patient's Global Impression of Change (PGIC) at Month 1 | Baseline and Month 1
  The change of overall health condition is assessed by PGIC and compared with baseline PGIC score. PGIC score has a minimum of 1 and a maximum of 7. Higher scores mean a greater improvement in health condition.
Global impression: Change From Baseline in Patient's Global Impression of Change (PGIC) at Month 3 | Baseline and Month 3
  The change of overall health condition is assessed by PGIC and compared with baseline PGIC score. PGIC score has a minimum of 1 and a maximum of 7. Higher scores mean a greater improvement in health condition.
Global impression: Change From Baseline in Patient's Global Impression of Change (PGIC) at Month 6 | Baseline and Month 6
  The change of overall health condition is assessed by PGIC and compared with baseline PGIC score. PGIC score has a minimum of 1 and a maximum of 7. Higher scores mean a greater improvement in health condition.
Global impression: Change From Baseline in Clinical Global Impressions-Improvement (CGI-I) at Month 1 | Baseline and Month 1
  The change of overall health condition is assessed by physicians using the CGI-I and compared with baseline CGI-I score. CGI-I score has a minimum of 1 and a maximum of 7. Higher scores mean a greater improvement in health condition.
Global impression: Change From Baseline in Clinical Global Impressions-Improvement (CGI-I) at Month 3 | Baseline and Month 3
  The change of overall health condition is assessed by physicians using the CGI-I and compared with baseline CGI-I score. CGI-I score has a minimum of 1 and a maximum of 7. Higher scores mean a greater improvement in health condition.
Global impression: Change From Baseline in Clinical Global Impressions-Improvement (CGI-I) at Month 6 | Baseline and Month 6
  The change of overall health condition is assessed by physicians using the CGI-I and compared with baseline CGI-I score. CGI-I score has a minimum of 1 and a maximum of 7. Higher scores mean a greater improvement in health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lu, MD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han Y, Lu Y, Wang D, Ran M, Ren Q, Xie D, Aziz TZ, Li L, Wang JJ. The Use of Remote Programming for Spinal Cord Stimulation for Patients With Chronic Pain During the COVID-19 Outbreak in China. Neuromodulation. 2021 Apr;24(3):441-447. doi: 10.1111/ner.13382. Epub 2021 Mar 22. PMID 33751731
- [Background] Lu Y, Xie D, Zhang X, Dong S, Zhang H, Yu B, Wang G, Wang JJ, Li L. Management of Intractable Pain in Patients With Implanted Spinal Cord Stimulation Devices During the COVID-19 Pandemic Using a Remote and Wireless Programming System. Front Neurosci. 2020 Dec 8;14:594696. doi: 10.3389/fnins.2020.594696. eCollection 2020. PMID 33363453
- [Derived] Cheng Y, Xie D, Han Y, Guo S, Sun Z, Jing L, Man W, Liu D, Yang K, Lei D, Meng Z, Zhang H, Wang G, Wu W, Wang G, Lu Y. Precise management system for chronic intractable pain patients implanted with spinal cord stimulation based on a remote programming platform: study protocol for a randomized controlled trial (PreMaSy study). Trials. 2023 Sep 11;24(1):580. doi: 10.1186/s13063-023-07595-4. PMID 37691092